CLINICAL TRIAL: NCT01782833
Title: A Prospective, Post Marketing Observational Study to Evaluate the Safety of Pletaal® SR Capsule
Brief Title: Pletaal SR Post Marketing Observational Study
Acronym: PLTSRPMOS
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 021-KOA-1201n
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Symptoms; Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: This is Non-interventional study

SUMMARY:
This is a Post Marketing Observational Study of cilostazol (Pletaal® SR capsule). As this study is observational in nature to collect the safety data after administrating the Pletaal SR capsule, from baseline to 16 weeks.

DETAILED DESCRIPTION:
This study will be conducted in a prospective, single-arm, multi-center format. As this study is observational in nature, the patient's follow-up is not prescriptive in nature and must be left up to the judgment of the physician (investigator), within the period of observation set forth in the protocol.

ELIGIBILITY:
Inclusion Criteria:

- Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study : 1. Patients who are prescribed Pletaal® SR capsule treatment as per investigator's medical judgment for adults aged 19 and over.

2. Patients who gave written authorization to use their personal and health data Physician (Investigator) will refer to the product market authorization (package insert) for inclusion criteria.

Exclusion Criteria:

* Patients presenting with any of the following will not be included in the study 1. Patients with hemorrhage 2. Patients with congestive heart failure 3. Patients with known hypersensitivity to Cilostazole or any ingredients of Pletaal® 4. Women who are pregnant or may possibly become pregnant 5. Patients who is not eligible to participate this study as investigator's medical judgment Physician (Investigator) will refer to the product market authorization (package insert) for exclusion criteria.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient who has below indication (1. Treatment of ischemic symptoms including ulceration, pain and coldness in chronic arterial occlusion (Berger's disease, arteriosclerosis obliterans, diabetic peripheral angiopathy). 2. Prevention of recurrence of cerebral infarction (excluding cardiogenic cerebral embolism).)
Sampling Method: Probability Sample
Enrollment: 3635 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - NHIC Ilsan Hospital, Goyang
  - Inje University Seoul Pail Hospital, Seoul
  - Seoul National University, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Pletaal® SR Capsule: Patients who were receiving or planned to receive Pletaal® SR Capsule according to investigator's medical judgement after a written contract with the study site and provided a written consent to use personal information.
Period: Overall Study
Arm/Group | Pletaal® SR Capsule
Started | 3635
Completed | 3365
Not Completed | 270

BASELINE CHARACTERISTICS:
Groups:
- Pletaal® SR Capsule: Subjects who received at least 1 dose of Pletaal® SR Capsule during the study period and had follow-up for safety assessment.
Arm/Group | Pletaal® SR Capsule
Number analyzed (Participants) | 3365
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.27 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1920
  Male | 1445

OUTCOME MEASURES:

1. Primary Outcome: The Incidence Rate and the Number of AE/ADRs
Description: Incidence rates of overall AEs and ADRs that occurred during the study period
Time Frame: Follow-up at least once from baseline to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pletaal® SR Capsule
Number analyzed (Participants) | 3365
Participants
  Number of patients reported for AE | 446
  Number of patients reported for ADR | 155

2. Secondary Outcome: The Incidence Rate of Tarchycardia and Palpitation After Pletaal® SR Capsule Administration
Time Frame: Follow-up at least once from baseline to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pletaal® SR Capsule
Number analyzed (Participants) | 3365
Participants
  Number of patients reported for 'Tachycardia' | 5
  Number of patients reported for 'Palpitat | 19

3. Secondary Outcome: The Number and Percentage of Drop-out Patients According to Aes
Time Frame: Follow-up at least once from baseline to 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pletaal® SR Capsule
Number analyzed (Participants) | 3365
Participants | 147

ADVERSE EVENTS:
Arm/Group | Pletaal® SR Capsule
Serious Adverse Events (participants affected / at risk) | 74/3365
Other Adverse Events (participants affected / at risk) | 372/3365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pletaal® SR Capsule (N=3365)
Cerebral infarction (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Central pain syndrome (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Intracranial artery dissection (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Cellulitis (Infections and infestations) | 1 (1)
Lung abscess (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Pyometra (Infections and infestations) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Oedema (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (General disorders) | 1 (1)
Cholelithiasis obstructive (General disorders) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Intraocular lens implant (Surgical and medical procedures) | 1 (1)
Peritoneal dialysis (Surgical and medical procedures) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2)
Diabetic vascular disorder (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pletaal® SR Capsule (N=3365)
Headache (Nervous system disorders) | 91 (91)
Dizziness (Nervous system disorders) | 42 (42)
Paraesthesia (Nervous system disorders) | 8 (8)
Hypoaesthesia (Nervous system disorders) | 7 (7)
Cerebral infarction (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 3 (3)
Amnesia (Nervous system disorders) | 2 (2)
Dizziness postural (Nervous system disorders) | 2 (2)
Hemiparesis (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Cerebellar ataxia (Nervous system disorders) | 1 (1)
Cervicogenic headache (Nervous system disorders) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Resting tremor (Nervous system disorders) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 17 (17)
Dyspepsia (Gastrointestinal disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Epigastric discomfort (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 2 (2)
Melaena (Gastrointestinal disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Oedema (General disorders) | 9 (9)
Chest pain (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 4 (4)
Chest discomfort (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Asthenia (General disorders) | 1 (1)
Face oedema (General disorders) | 2 (2)
General symptom (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Localised oedema (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Periodontitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1)
Palpitations (Cardiac disorders) | 19 (19)
Tachycardia (Cardiac disorders) | 5 (5)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Chloasma (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Blood glucose increased (Investigations) | 4 (4)
Liver function test abnormal (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bacterial test (Investigations) | 1 (1)
Blood glucose abnormal (Investigations) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Lipids increased (Investigations) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1)
Urobilinogen urine increased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7)
Anxiety (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Dysthymic disorder (Psychiatric disorders) | 1 (1)
Hallucination, auditory (Psychiatric disorders) | 1 (1)
Mood altered (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 3 (3)
Otorrhoea (Ear and labyrinth disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Peripheral coldness (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Flushing (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Diabetic retinopathy (Eye disorders) | 1 (1)
Dacryostenosis acquired (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 2 (2)
Polypectomy (Surgical and medical procedures) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol (2012-07-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT01782833/Prot_000.pdf